CLINICAL TRIAL: NCT01350323
Title: Aqueous Humor Levels of Vascular Endothelial Growth Factor Before and After Intravitreal Bevacizumab in Type 3 Versus Type 1 and 2 Neovascularization. A Prospective, Case-control Study.
Brief Title: Aqueous Vascular Endothelial Growth Factor (VEGF) Levels in Type 3 Neovascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Roberto dell'Omo, University of Molise
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: UM-O-1
Record Dates: First submitted 2011-05-02; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2009-03

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Type 3 NV (Active Comparator): Wet-AMD related type 3 neovascularization
  Interventions: Procedure: Aqueous sample
- Type 2 NV (Active Comparator): Wet-AMD related type 2 neovascularization
  Interventions: Procedure: Aqueous sample
- Type 1 NV (Active Comparator): Wet-AMD related type 1 neovascularization
  Interventions: Procedure: Aqueous sample
- Controls (Other): Aqueous sample (0.1ml) in patients undergoing cataract extraction
  Interventions: Procedure: Aqueous sample

INTERVENTIONS:
Procedure: Aqueous sample — Aqueous sample (0.1ml of aqueous)+ intravitreal injection of bevacizumab (1.25mg/0.05ml)
  Other Names: Avastin
  Arms: Type 3 NV
Procedure: Aqueous sample — Aqueous sample (0.1ml)+intravitreal injection of bevacizumab (1.25mg/0.05ml)
  Other Names: Avastin
  Arms: Type 2 NV
Procedure: Aqueous sample — Aqueous sample (0.1ml)+ intravitreal injection of bevacizumab (1.25mg/0.05ml)
  Other Names: Avastin
  Arms: Type 1 NV
Procedure: Aqueous sample — Aqueous sample (0.1ml)
  Other Names: Avastin
  Arms: Controls

SUMMARY:
This is a pilot, prospective, interventional, case-control study investigating aqueous levels of vascular endothelial growth factor (VEGF) in eyes with AMD-related neovascularization treated with intravitreal bevacizumab at the Medical Retina Department, University of Molise, Campobasso.

DETAILED DESCRIPTION:
This was a pilot, prospective, interventional, case-control study investigating aqueous levels of VEGF in eyes with AMD-related NV treated with intravitreal bevacizumab.

Classification of neovascularization was based on its anatomic localization as ascertained by multimodal imaging employing FA (fluorescein angiography), ICGA (indocyanine green angiography) and OCT (optical coherence tomography) as recently proposed by Freund et al.

Diagnostic procedures and follow-up At baseline all the patients underwent BCVA measurement using early treatment diabetic retinopathy study (ETDRS) chart at 4 meters, fundus biomicroscopy, FA, ICGA and sd-OCT. All examinations were repeated in occasion of the follow-up appointments with exception of angiographic tests.

Angiographic tests and OCTs scans were recorded using Spectralis sd-OCT (Spectralis SD-OCT, Heidelberg Engineering, Heidelberg, Germany).

CMT was calculated after acquiring a sequence of 145 horizontal sections recorded in the high-resolution mode (1024 A-scans/30 degrees) and covering an area of 20 degrees (horizontal) × 15 degrees (vertical) with a distance of ~30 µm between individual sections. On follow-up examinations, the imaging processing software allowed reevaluation at exactly the same location.

The images were then processed by the "Thickness Map" analysis program. Field 1 of the map analysis protocol (central 1 mm) was used for central retinal thickness calculations.

Aqueous Sampling and Bevacizumab Injections All patients with AMD-related neovascularization received three intravitreal injections of 1.25 mg/0.05 ml of bevacizumab (Avastin; Genentech Inc, South San Francisco, California, USA) at baseline, month 1 and month 2.

Before injection, topical anesthesia was induced by tetracaine (1%) eye drops. Povidone-iodine was applied to the eyelid margins, the lashes, the conjunctiva bulbi and the fornices. After application of a sterile drape, a lid speculum was inserted.

Immediately before each intravitreal injection, aqueous sampling was performed by aspirating 0.05-0.1 ml of aqueous using a 30-gauge needle connected to a tuberculin syringe at the temporal limbus. All the samples were collected in the operating theatre under operating microscope control.

Intravitreal bevacizumab (IVB) injection was then performed using a 30-gauge needle in the inferotemporal quadrant at 3.5 mm to 4 mm posterior to the limbus.

The undiluted aqueous samples were transferred into sterile containers and immediately stored in a -80°C freezer until analysis.

Control Group Reference samples were obtained from 14 age-matched patients undergoing cataract surgery.

Aqueous humor samples were obtained in the same fashion described above for eyes with wet-AMD. The undiluted aqueous samples were transferred into sterile containers and immediately stored in a -80°C freezer until analysis.

Vascular Endothelial Growth Factor Assay Collected samples were gradually equilibrated to room temperature before beginning the assay and diluted 1:1 with the sample diluent provided by the manufacturer.

The VEGF content was determined on 50 µl of diluted sample with a human VEGF ELISA kit (EHVEGF, Pierce Biotechnology, Rockford, Illinois, USA) according to the manufacturer's instruction and using an extended standard curve including a 16, 8 and 4 pg/ml standard point. All assays were performed in duplicate. The minimum detectable concentration of VEGF was 3.5 pg/ml. Values inferior to 3.5pg/ml were considered equal to 1 for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* wet age-related macular degeneration type 1, 2 or 3

Exclusion Criteria:

* BCVA at baseline less than 1.0 logMAR
* any previous treatment of the neovascular lesion
* previous vitrectomy
* laser coagulation within the last 3 months
* previous participation in any studies using investigational drugs within 3months preceding day 0
* intraocular surgery (including cataract surgery) in the study eye within 3 months preceding day 0
* glaucoma in the study eye; diabetes mellitus
* use of immunosuppressive drugs
* malignant tumors of any location

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Aqueous VEGF concentration | Change from baseline of VEGF concentration at month 1
  To establish if different types of wet-AMD were associated to different concentrations of VEGF at baseline

SECONDARY OUTCOMES:
Macular thickness assessment | Change from baseline of macular thickness at month 1
  to compare central macular thickness before and after treatment respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto dell'Omo, MD, Principal Investigator — University of Molise; Ciro Costagliola, Professor, Study Director — University of Molise
Locations (1):
- University of Molise, Campobasso, Italy

REFERENCES:
- [Background] Yannuzzi LA, Negrao S, Iida T, Carvalho C, Rodriguez-Coleman H, Slakter J, Freund KB, Sorenson J, Orlock D, Borodoker N. Retinal angiomatous proliferation in age-related macular degeneration. Retina. 2001;21(5):416-34. doi: 10.1097/00006982-200110000-00003. PMID 11642370
- [Background] Bottoni F, Massacesi A, Cigada M, Viola F, Musicco I, Staurenghi G. Treatment of retinal angiomatous proliferation in age-related macular degeneration: a series of 104 cases of retinal angiomatous proliferation. Arch Ophthalmol. 2005 Dec;123(12):1644-50. doi: 10.1001/archopht.123.12.1644. PMID 16344434
- [Background] Wells JA, Murthy R, Chibber R, Nunn A, Molinatti PA, Kohner EM, Gregor ZJ. Levels of vascular endothelial growth factor are elevated in the vitreous of patients with subretinal neovascularisation. Br J Ophthalmol. 1996 Apr;80(4):363-6. doi: 10.1136/bjo.80.4.363. PMID 8703891